CLINICAL TRIAL: NCT05639439
Title: Comparative Evaluation of Periglottic Airway Devices With Performed Shape
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Evanthia Dimitriou, Anesthesiologist, MD, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12/03/2021anesthesia
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Airway Management
Keywords: ventilation; airway management; periglottic airway device
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A- Fastrach (Active Comparator): Group of 40 patients scheduled for elective surgery under general anesthesia are planned to be ventilated through the intubating laryngeal mask airway "Fastrach", while the laryngeal view through "Fastrach" will be evaluated using a flexible fiberoptic bronchoscope
  Interventions: Device: Ventilation using the "Fastrach" intubating laryngeal mask airway and glottic view using fibrescope - Group A
- Group B- Proseal (Active Comparator): Group of 40 patients scheduled for elective surgery under general anesthesia are planned to be ventilated through the "Proseal" laryngeal mask airway, while the laryngeal view through "Proseal" will be evaluated using a flexible fiberoptic bronchoscope
  Interventions: Device: Ventilation using the "Proseal" laryngeal mask airway and glottic view using fibrescope- Group B
- Group C- I-gel (Active Comparator): Group of 40 patients scheduled for elective surgery under general anesthesia are planned to be ventilated using the "I-gel" supraglottic airway device, while the laryngeal view through "I-gel" will be evaluated using a flexible fiberoptic bronchoscope
  Interventions: Device: Ventilation using the "I-gel" supraglottic airway device and glottic view using fibrescope- Group C
- Group D- Protector (Active Comparator): Group of 40 patients scheduled for elective surgery under general anesthesia are planned to be ventilated using the "Protector" laryngeal mask airway, while the laryngeal view through "Protector" will be evaluated using a flexible fiberoptic bronchoscope
  Interventions: Device: Ventilation using the "Protector" laryngeal airway device and glottic view using fibrescope- Group D

INTERVENTIONS:
Device: Ventilation using the "Fastrach" intubating laryngeal mask airway and glottic view using fibrescope - Group A — Insertion of the intubating laryngeal airway device "Fastrach", evaluation of the ventilation sufficiency and perfection of installation/ anatomical application to the larynx (evaluation with fiberoptic bronchoscope)
  Arms: Group A- Fastrach
Device: Ventilation using the "Proseal" laryngeal mask airway and glottic view using fibrescope- Group B — Insertion of the laryngeal airway device "Proseal", evaluation of the ventilation sufficiency and perfection of installation/ anatomical application to the larynx (evaluation with fiberoptic bronchoscope)
  Arms: Group B- Proseal
Device: Ventilation using the "I-gel" supraglottic airway device and glottic view using fibrescope- Group C — Insertion of the supraglottic airway device "I-gel", evaluation of the ventilation sufficiency and perfection of installation/ anatomical application to the larynx (evaluation with fiberoptic bronchoscope)
  Arms: Group C- I-gel
Device: Ventilation using the "Protector" laryngeal airway device and glottic view using fibrescope- Group D — Insertion of the laryngeal airway device "Protector", evaluation of the ventilation sufficiency and perfection of installation/ anatomical application to the larynx (evaluation with fiberoptic bronchoscope)
  Arms: Group D- Protector

SUMMARY:
The purpose of this study is to evaluate four, most popular periglottic airway devices as regards to ventilation sufficiency and perfection of installation/ anatomical application to the larynx (evaluation with fiberscope).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients (>18 years old scheduled for elective surgery under general anesthesia) giving written informed consent will undergo preoperative screening examination to determine eligibility for study entry. A randomization process has been previously done, according to which the participants have been classified into one of the four groups of the study. Each study group is scheduled to receive one of the four periglottic devices (LM FastrachTM, LM ProsealTM, LM I-GelTM, LM ProtectorTM) while evaluating the ventilation sufficiency and perfection of installation/ anatomical application to the larynx (evaluation with fiberscope).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old, undergoing elective surgery under general anesthesia

Exclusion Criteria:

* Patients < 18 years old
* Patients undergoing emergency surgery or trauma patients
* Obstetric population
* Patients receiving regional anesthesia
* Patients to whom the use of periglottic airway device is contraindicated
* Patients with RODS score ≥ 1 (score to predict difficult laryngeal mask placement 1-4)
* Patients with anticipated difficult airway, planned for awake intubation
* Patients' refusal to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Ventilation sufficiency | Up to study completion, an average of 2 years
  Evaluation of ventilation sufficiency using manual bag-periglottic airway device ventilation (sufficient- moderate sufficient- insufficient)
Time required for successful periglottic airway device placement | Up to study completion, an average of 2 years
  Time required from the beginning of the insertion of the periglottic airway device until the appearance of the first capnographic waveform with end-tidal CO2> 20mmHg
Perfection of installation/ anatomical application to the larynx | Up to study completion, an average of 2 years
  After sufficient placement of the periglottic devise, a fibrescope is inserted through the mask in order to evaluate the glottic view (grade I-IV) and the anatomical application of the mask to the larynx.

SECONDARY OUTCOMES:
Leak pressure | Up to study completion, an average of 2 years
  The leak pressure of each mask will be measured applying fresh gas flow (FGF) of 3L/min while keeping the adjustable pressure- limiting (APL) valve closed.

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Dimitriou, MD, Principal Investigator — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Pátrai, Ahaia, Greece